CLINICAL TRIAL: NCT02042833
Title: An Observational Study of Patients' Perception of Treatment With Erythropoiesis-Stimulating Agents in Patients With Chronic Kidney Disease Not on Dialysis (PERCEPOLIS)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25557
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate patients' perception of treatment with erythropoiesis-stimulating agents in patients with chronic kidney disease not on dialysis. Eligible patients initiated on treatment with Mircera (methoxy polyethylene glycol-epoetin beta) will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients with chronic kidney disease not on dialysis (with or without previous renal transplantation)
* Treated or not with ESA at time of visit
* Patients for whom the treating physician had decided to initiate Mircera for medical reasons before the commencement of the study
* Initiation of treatment with Mircera at the inclusion visit
* Accepting and able of completing the ESA preference questionnaire

Exclusion Criteria:

* Participation in a clinical trial on anemia
* Treatment with Mircera during the 3 months before inclusion
* Dialysis planned in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease not on dialysis (with or without previous renal transplantation), initiating treatment with Mircera, and erythropoiesis-stimulating agent (ESA)-naïve or not
Sampling Method: Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Relative importance for patients of different attributes of ESA treatment, assessed by Choice Based Conjoint questionnaire at baseline and Month 6 | 6 months

SECONDARY OUTCOMES:
Biological parameters: hemoglobin concentration at each observation time point. | 6 months
Adherence to Mircera treatment assessed by a questionnaire adapted from the Morisky scale at baseline and at Month 6 | 6 months
Dose/schedule of Mircera treatment at each observation timepoint | 6 months
Concomitant medication/treatments in the management of anemia | 6 months
Proportion of patients with a hemoglobin level between 10 and 12 g/dL after 6 months of treatment with Mircera | Month 6
Change in hemoglobin level | from baseline to Month 6
Safety: Incidence of adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (92):
- France (92):
  - Aix-en-Provence
  - Ajaccio
  - Annonay
  - Arras
  - Avignon
  - Bagnols-sur-Cèze
  - Bayonne
  - Beauvais
  - Belley
  - Besançon
  - Bièvres
  - Bois-Guillaume
  - Bordeaux
  - Bourg-en-Bresse
  - Bourgoin
  - Brest
  - Cabestany
  - Caen
  - Castelnau-le-Lez
  - Chalon-sur-Saône
  - Champigny-sur-Marne
  - Charleville-Mézières
  - Chaumont
  - Châteauroux
  - Clermont-Ferrand
  - Colmar
  - Creil
  - Créteil
  - Dijon
  - Dole
  - Draguignan
  - Épinal
  - Évian-les-Bains
  - Évreux
  - Freyming-Merlebach
  - Gap
  - Gradignan
  - Greize
  - Grenoble
  - Haguenau
  - La Chaussée-Saint-Victor
  - La Roche-sur-Yon
  - La Tronche
  - Laon
  - Le Mans
  - Le Puy-en-Velay
  - Lille
  - Lorient
  - Lyon
  - Marseille
  - Maubeuge
  - Mâcon
  - Melun
  - Metz
  - Mont-de-Marsan
  - Mont-Saint-Martin
  - Montluçon
  - Mullhouse
  - Nancy
  - Nantes
  - Nice
  - Nîmes
  - Olivet
  - Ollioules
  - Orléans
  - Paris
  - Perpignan
  - Pierre-Bénite
  - Poissy
  - Poitiers
  - Quimper
  - Rambouillet
  - Rennes
  - Roanne
  - Rodez
  - Romans-sur-Isère
  - Rouen
  - Saint-Laurent-du-Var
  - Saint-Lô
  - Saint-Priest-en-Jarez
  - Saint-Quentin
  - Salouël
  - Sens
  - Strasbourg
  - Toulon
  - Toulouse
  - Tournan-en-Brie
  - Tours
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vannes
  - Vesoul